CLINICAL TRIAL: NCT00620035
Title: An Open-Label, Non-Controlled Multicenter Trial to Evaluate the Insertion Characteristics of the Radiopaque Etonogestrel Implant Using a Next Generation Applicator
Brief Title: A Multicenter Trial to Evaluate the Insertion Characteristics of the Radiopaque Etonogestrel Implant Using a Next Generation Applicator (34530)(P05702)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: P05702; 34530
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2011-10-31 (Estimated); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiopaque Etonogestrel Implant (Experimental): Radiopaque Etonogestrel Implant (drug) inserted with the Next Generation Applicator (NGA)
  The Radiopaque Implant is a single rod contraceptive implant of 4 cm length and
  2 mm in diameter which is placed at the inner side of the non-dominant upper-arm
  about 8-10 cm above the medial epicondyle. The Radiopaque Implant contains
  approximately 68 mg etonogestrel (ENG) dispersed in a matrix of ethylene vinyl acetate (EVA) copolymer and barium sulfate, surrounded by an EVA membrane. The barium-sulfate provides radio-opacity and allows detection by X-ray.
  The ENG dose released from the implant amounts to about 60-70 mcg/day shortly after insertion and decreases to about 40 mcg/day at the start of the second year, and to about 25-30 mcg/day at the end of the third year.
  Interventions: Drug: Radiopaque Etonogestrel Implant

INTERVENTIONS:
Drug: Radiopaque Etonogestrel Implant — One implant inserted for a 3-year treatment period
  Other Names: SCH 900415

SUMMARY:
The primary purpose of this study is to evaluate the use of the next generation applicator and its instructions for proper insertion of the Radiopaque Implant. Secondary objectives include: evaluation of implant removal, evaluation of the overall contraceptive efficacy and safety of the Radiopaque Implant, assessment of x -ray visibility of the Radiopaque Implant, and to assess participant expectations and satisfaction with the Radiopaque Implant.

ELIGIBILITY:
Inclusion Criteria:

* Woman of at least (>=) 18 but not older than (<= )40 years of age at the time of screening;
* Good physical and mental health;
* Regular cycles with a usual length between 24 and 35 days;
* Body mass index >= 18 and <= 35 kg/m^2;
* Willing to give informed consent in writing.

Exclusion Criteria:

* Contraindications:

  * known or suspected pregnancy;
  * active venous thromboembolic disorder (e.g. deep vein thrombosis,

pulmonary embolism);

* presence or history of severe hepatic disease as long as liver function values have not returned to normal;
* malignancy or pre-malignancy, if sex-steroid-influenced;
* undiagnosed vaginal bleeding;
* hypersensitivity to any of the components of Radiopaque Implant.

  * Hypertension, i.e. systolic blood pressure >140 mmHg and/or diastolic blood pressure > 90 mmHg;
  * A history during pregnancy or during previous use of sex steroids of: jaundice and/or severe pruritus related to cholestasis, gallstone formation, porphyria, systemic lupus erythematosus, haemolytic uraemic syndrome, Sydenham's chorea, herpes gestationis, otosclerosis-related hearing loss;
  * Present use or use during 2 months prior to the start of Radiopaque Implant of one of the following drugs: phenytoin, phenobarbital, primidone, carbamazepine, rifampicin, oxcarbazepine, topiramate, felbamate, ritonavir, nelfinavir, griseofulvin or the herbal remedy St John's wort;
  * Administration of investigational drugs within 2 months prior to the start of Radiopaque Implant

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

REFERENCES:
- [Derived] Mommers E, Blum GF, Gent TG, Peters KP, Sordal TS, Marintcheva-Petrova M. Nexplanon, a radiopaque etonogestrel implant in combination with a next-generation applicator: 3-year results of a noncomparative multicenter trial. Am J Obstet Gynecol. 2012 Nov;207(5):388.e1-6. doi: 10.1016/j.ajog.2012.08.002. Epub 2012 Aug 10. PMID 22939402

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At screening, a participant number was allocated to 308 participants of which 7 participants did not receive treatment. A total of 301 participants had an implant inserted.
Groups:
- Radiopaque Etonogestrel Implant: The Radiopaque Implant is a single rod contraceptive implant of 4 cm length and 2 mm in diameter which is placed at the inner side of the non-dominant upper-arm about 8-10 cm above the medial epicondyle. The Radiopaque Implant contains approximately 68 mg etonogestrel (ENG) dispersed in a matrix of ethylene vinyl acetate (EVA) copolymer and barium sulfate, surrounded by an EVA membrane. The barium-sulfate provides radio-opacity and allows detection by X-ray.
  The ENG dose released from the implant amounts to about 60-70 mcg/day shortly after insertion and decreases to about 40 mcg/day at the start of the second year, and to about 25-30 mcg/day at the end of the third year.
Period: Overall Study
Arm/Group | Radiopaque Etonogestrel Implant
Started | 301
Completed | 156
Not Completed | 145
Not completed — Adverse Event | 106
Not completed — Withdrawal of Informed Consent | 1
Not completed — Other Reason | 38

BASELINE CHARACTERISTICS:
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 301
Age, Customized [Number; unit: participants]
  18-20 years | 43
  21-25 years | 79
  26-30 years | 64
  31-35 years | 54
  36-40 years | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 301
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Applicator Users Who Were Very Satisfied and Satisfied- User Satisfaction Questionnaire for Domain: Design & Technical Aspects
Description: In order to evaluate efficacy and ease of use of the Next Generation Applicator (NGA), the investigator/applicator user (AU) completed a User Satisfaction Questionnaire on Day 1 after the 12th implant insertion. The domain, 'Design/technical aspects' consisted of five questions: fit of the applicator in the hand, size, weight, handling, and color of the applicator were assessed. The percentage of AUs who were very satisfied and satisfied was presented.
Time Frame: Day 1
Population: The Applicator User (AU) group consisted of all investigators participating in the trial and who performed at least one insertion.
Measure: Number; unit: Percentage of Applicator Users
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 23
Percentage of Applicator Users | 99.1

2. Primary Outcome: Percentage of Applicator Users Who Were Very Satisfied and Satisfied- User Satisfaction Questionnaire for Domain: Functionality
Description: In order to evaluate efficacy and ease of use of the NGA, the investigator/AU completed a User Satisfaction Questionnaire on Day 1 after the 12th implant insertion. The domain, 'Functionality' consisted of six questions assessing functionality of the needle. The percentage of AUs who were very satisfied and satisfied was presented.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Applicator Users
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 23
Percentage of Applicator Users | 94.9

3. Primary Outcome: Percentage of Applicator Users Who Were Very Satisfied and Satisfied- User Satisfaction Questionnaire by Domain: Safety
Description: In order to evaluate efficacy and ease of use of the NGA, the investigator/AU completed a User Satisfaction Questionnaire on Day 1 after the 12th implant insertion. The domain, 'Safety' consisted of three questions: removal of the protection cap from applicator, full retraction of the needle into the applicator after insertion, difference in colors of the obturator & the implant. The percentage of AUs who were very satisfied and satisfied was presented.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Applicator Users
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 23
Percentage of Applicator Users | 98.6

4. Primary Outcome: Percentage of Applicator Users Who Were Very Satisfied and Satisfied- User Satisfaction Questionnaire for Domain: Used Time
Description: In order to evaluate efficacy and ease of use of the NGA, the investigator/AU completed a User Satisfaction Questionnaire on Day 1 after the 12th implant insertion. The domain, 'Used Time' consisted of one question: insertion time was assessed. The percentage of AUs who were very satisfied and satisfied was presented.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Applicator Users
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 23
Percentage of Applicator Users | 100

5. Primary Outcome: Percentage of Applicator Users Who Were Very Satisfied and Satisfied- User Satisfaction Questionnaire for Domain: Applicator Satisfaction
Description: In order to evaluate efficacy and ease of use of the NGA, the investigator/AU completed a User Satisfaction Questionnaire on Day 1 after the 12th implant insertion. The domain, 'Applicator Satisfaction' consisted of one question in order to assess the applicator. The percentage of AUs who were very satisfied and satisfied was presented.
Time Frame: Day 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Applicator Users
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 23
Percentage of Applicator Users | 100

6. Primary Outcome: Implant Insertion Time (Seconds)
Description: The implant insertion time was the time expressed in seconds, from removal of the protection cap from the applicator until retraction of the needle from the arm after insertion. Data was presented for overall investigators including experienced and non-experienced.
Time Frame: Day 1
Population: All-Subjects-Treated (AST) group included all participants who had the Radiopaque implant inserted (N=301). Data was reported for 291 implant insertions.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 291
Seconds | 27.9 (29.3)

7. Primary Outcome: Implant Removal Time (Seconds)
Description: The implant removal time was the time expressed in seconds, from making the removal incision until placing the butterfly closure. Data was presented for overall investigators including experienced and non-experienced.
Time Frame: Day 1
Population: All-Subjects-Treated (AST) group included all participants who had the Radiopaque implant inserted (N=301). Data was reported for 292 implant removals.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Radiopaque Etonogestrel Implant
Number analyzed (Participants) | 292
Seconds | 119.3 (120.2)

ADVERSE EVENTS:
Time Frame: Safety data from the actual in-treatment period was used. The in-treatment period started on the day of the implant insertion and continued up to and including the fifth day after implant removal (3 years).
Description: The safety analysis was performed for the AST group; all subjects who had the Radiopaque Implant inserted.
Arm/Group | Radiopaque Etonogestrel Implant
Serious Adverse Events (participants affected / at risk) | 17/301
Other Adverse Events (participants affected / at risk) | 233/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiopaque Etonogestrel Implant (N=301)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1)
Salpingo-oophoritis (Infections and infestations) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Bipolar Disorder (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 1 (1)
Calculus Urinary (Renal and urinary disorders) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiopaque Etonogestrel Implant (N=301)
Implant Site Haematoma (General disorders) | 16 (16)
Implant Site Pain (General disorders) | 18 (20)
Influenza (Infections and infestations) | 19 (22)
Nasopharyngitis (Infections and infestations) | 32 (45)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (30)
Urinary Tract Infection (Infections and infestations) | 20 (31)
Vulvovaginal Candidiasis (Infections and infestations) | 19 (26)
Weight Increased (Investigations) | 35 (38)
Headache (Nervous system disorders) | 56 (103)
Amenorrhoea (Reproductive system and breast disorders) | 21 (23)
Dysmenorrhoea (Reproductive system and breast disorders) | 16 (18)
Menorrhagia (Reproductive system and breast disorders) | 31 (35)
Metrorrhagia (Reproductive system and breast disorders) | 53 (60)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 85 (126)
Acne (Reproductive system and breast disorders) | 39 (48)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR recognizes the right of the investigator(s) to publish, but all publications must be based on data validated and released by SPONSOR. Any such scientific paper, presentation, or other communication concerning the clinical trial described in protocol will first be submitted to SPONSOR, at least six weeks ahead of estimated publication or presentation, for written consent, which shall not be withheld unreasonably.